CLINICAL TRIAL: NCT05541419
Title: Efficacy of Addition of High-volume Nasal Wash With Budesonide Diluted to Maximum Clinical Treatment of Patients With Chronic Rhinosinusitis With Polyoposis: Double, Randomized, Controlled Double Study
Brief Title: Use of Budesonide Diluted to Maximum Clinical Treatment of Patients With Chronic Rhinosinusitis With Polyoposis.
Acronym: CRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Marco Aurélio Fornazieri, Principal Investigator, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFornazieri
Record Dates: First submitted 2022-08-24; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Rhinosinusitis; Quality of life
MeSH Terms: conditions — Disease; Rhinosinusitis | interventions — Placebo Effect

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maximum clinical treatment + Budesonide diluted (Experimental): The maximum clinical treatment consists of intramuscular injection of Dispropan® in intramuscular injectable suspension and busonid in nasal spray, two sprays of 50mcg in each nostril.
  In this study, the investigator wishes to add to the maximum clinical treatment a daily wash with high volume diluted budesonide.
  Interventions: Drug: Budesonide Nasal
- Maximum clinical treatment + Placebo (Placebo Comparator): To compare the efficacy of adding diluted budesonide lavage to maximal clinical treatment, the placebo group is used. The placebo formula is composed of 1% glycerin diluted in water.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Budesonide Nasal — The patient performed a lavage once daily with 2mg dilute budesonide. The maximum clinical treatment consists of intramuscular injection of Dispropan® in intramuscular injectable suspension and busonid in nasal spray, two sprays of 50mcg in each nostril.
  Other Names: Busonid
  Arms: Maximum clinical treatment + Budesonide diluted
Drug: Placebos — Composed of 1% glycerin diluted in water. The maximum clinical treatment consists of intramuscular injection of Dispropan® in intramuscular injectable suspension and busonid in nasal spray, two sprays of 50mcg in each nostril.
  Other Names: placebo effect
  Arms: Maximum clinical treatment + Placebo

SUMMARY:
This is a double-blind, randomized, double-blind, randomized, double-blind, randomized block design with two intervention groups of 30 patients each. Patients not recruited at the otorhinolaryngology outpatient clinic of the Regional University Hospital of the North of Paraná and the University Hospital Specialties Ambulatory will be included in the study of chronic rhinosinusitis with polyposis are randomly divided with stratification for the presence of two groups of patients. 30 patients, with 9 asthmatics in each). Of the nasal nasal with 2mg budesonide diluted in high daily volume added to the corticosteroid injectable injectable and the topic for 16 weeks compared to placebo. The Polyp Score (NPS), Sono-Nasal Outcome Test-22 (SNOT-22), University of Pennsylvania Olfactory Identification Test (UPSIT), peak nasal inspiratory flow (PNIF), visual scales preoperative tomography, acoustic rhinometry, computerized rhinomanometry and nasal endoscopy before and after the treatments. Position Paper on Nasal Rhinosinusitis and Nasal Polyps 2012; A bilateral nasal pole score is 5 and a maximum of 8 for both nostrils (with less than a score of 2 for each nostril).

DETAILED DESCRIPTION:
INTRODUTION: According to the European Position Paper on Rhinosinusitis and Nasal Polyps 2012, chronic rhinosinusitis in adults can be defined as an inflammation of the nasal mucosa and paranasal sinuses lasting 12 weeks or more , associated or not with nasal polyposis. As to the origin of the polyps, these are typically related to the eosinophilic inflammation of the upper airways and result in obstructions in different degrees of the nasal cavities. Maximum clinical treatment - a combination of several classes of drugs to optimize therapy - often proves to be the first choice in the management of this disease. There is, however, no consensus on the composition or duration of maximal clinical treatment, and success rates are extremely variable. If there is no improvement in the condition, surgical treatment is usually instituted and, if necessary, supplemented with topical post-operative treatment. Recent studies have led to the perception that sprays and aerosols can not adequately reach the paranasal sinuses resulting in a better effect of the medication, if possible, such methods should be replaced by nasal cavity lavages using high volume solutions. OBJECTIVES: The present study aims to compare, through validated tests, the impact of the inclusion of nasal lavage with budesonide diluted in high volume in relation to placebo, in the improvement of the symptoms, signs, and quality of life of patients with chronic rhinosinusitis with polyposis. If effective, this therapy may decrease surgical indications and, consequently, health expenditures for the government. METHODOLOGY: Parallel, randomized, placebo-controlled, parallel type clinical trial. Patients with chronic rhinosinusitis with polyposis will be divided randomly with stratification for the presence of asthma in two groups (two blocks of 30 patients, 9 asthmatics each). It will evaluate the effectiveness of nasal lavage with 2mg budesonide diluted in high volume daily added to the initial systemic corticosteroid injectable and the topic for 16 weeks compared to placebo. EXPECTED RESULTS: It is expected that diluted budesonide improvement in the symptoms, signs, and quality of life of patients with chronic rhinosinusitis with polyposis.

ELIGIBILITY:
Inclusion Criteria:

1. A minimum nasal polyp score (NPS) of 5 of a maximum of 8 for both nostrils (with at least a score of 2 for each nostril).
2. Presence of at least two of the following symptoms prior to screening: nasal blockage / obstruction / congestion or rhinorrhea (anterior or posterior); facial / pressure pain; reduction or loss of smell.

Exclusion Criteria:

1. A patient under the age of 18, or over 55;
2. SNOT-22 with sum of less than 7;
3. Patients who have used drugs or therapies that interfere with the results of this clinical trial within 2 months prior to screening: treatment with immunosuppressants; anti-immunoglobulin and within two months prior to screening.
4. Initiation of allergen immunotherapy within 3 months prior to first consultation or plan to initiate therapy during the screening period or randomized treatment period;
5. Patients who underwent any nasal surgery;
6. Patients on anti-leukotrienes and antihistamines
7. Asthmatic patients will be excluded if: forced expiratory volume (FEV1) is 60% predicted or lower; an exacerbation requiring systemic (oral and / or parenteral) or hospitalization for more than 24 hours for the treatment of asthma has occurred within 3 months prior to screening; use of a dose greater than 1000 μg of inhaled fluticasone or equivalent;
8. Patients with a short life expectancy (less than 6 months);

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the improvement in the Nasal Polyp Score | 16 weeks
  To verify, from the change in the Nasal Polyp Score (NPS, range from 0 to 8, higher score indicates larger polyp size), the impact of maximum clinical treatment - intramuscular injection of Dispropan in intramuscular injectable suspension and budesonide in nasal spray, two sprays of 50 mcg in each nostril - plus high-volume diluted budesonide nasal lavage, compared to the same maximum clinical treatment plus high-flow placebo nasal lavage in patients with chronic rhinosinusitis with polyposis without previous nasal surgery for a period of 16 weeks.

SECONDARY OUTCOMES:
Improves olfactory ability through the University of Pennsylvania Smell Identification Test | 16 weeks
  UNIVERSITY OF PENNSYLVANIA SMELL IDENTIFICATION TEST (UPSIT) - This instrument consists of four cards of 10 odors, with one odor per page. The stimuli are embedded in plastic microcapsules present in a brown band at the bottom of each page. The examiner directs the person being examined to scrape this strip with a pencil, which causes the odor to be released. After that, the patient answers a multiple choice question to describe what the odor looks like. Based on the score obtained, the individual's olfactory function can be classified into normosmia, microsmia (mild, moderate and severe) and anosmia (Fornazieri et al., 2010). This test has been validated for the Brazilian population (Fornazieri et al., 2015).
Sino-Nasal Outcome Test - 22 (SNOT-22) | 16 weeks
  The Sino-Nasal Outcome Test - 22 consists of a questionnaire consisting of 22 questions that assess the severity of nasal symptoms reported by the patient on a scale from 0 to 5 in each question, with a score of 5 being the greatest discomfort to the patient. The questions that make up the SNOT-22 refer to rhinological, otological, facial symptoms (12 questions) and their impact on quality of life (10 questions), which cover sleep function and psychological impairment. The questionnaire, as a whole, includes symptoms such as the need to blow nose, sneezing, rhinorrhea, cough, posterior rhinorrhea, thick rhinorrhea, ear fullness, dizziness, otalgia, facial pain or pressure, difficulty initiating sleep, fatigue on awakening, reduced of productivity and concentration, frustration, sadness and irritability (Piccirillo, Merritt and Richards, 2002; Hopkins et al., 2009).
Analogic visual scale (VAS) | 16 weeks
  The visual analogue scale for chronic rhinosinusitis is used to assess the severity of symptoms and their impact on the patient's quality of life, based on the question: "How problematic are your symptoms of rhinosinusitis?". The patient should mark, on a 10 centimeter line graduated on a scale from zero to ten, the severity of the symptoms reported, with zero representing no discomfort, and ten representing the greatest possible discomfort (Fokkens, Lund and Mullol, 2007) (Bachert et al., 2016).
  The disease can be divided into:
  Mild = patient scores between 0 and 3; Moderate = patient scores between 3 and 7; Severe = patient scores between 7 and 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Aurelio Fornazieri, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No